CLINICAL TRIAL: NCT01144325
Title: Minimally Invasive Esophagectomy in Prone or Left Decubitus Position: A Prospective Randomized Clinical Trial From A Single Institution
Brief Title: Minimally Invasive Esophagectomy (MIE) in Prone Versus Left Decubitus Position
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Tan, Lijie MD / Associate Professor of Surgery, Division of Thoracic Surgery, Zhong Shan Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: ZSchest2010001; MIEFUDANU2010001 (Other: Zhong Shan Hospital, Fu Dan University)
Record Dates: First submitted 2010-05-26; First posted 2010-06-15 (Estimated); Last update posted 2011-03-08 (Estimated); Status verified 2011-02

CONDITIONS: Esophageal Cancer; Esophagectomy
Keywords: Minimally Invasive Esophagectomy
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: thoracoscopic esophagectomy — In prone position group, patients are intubated with single lumen endotracheal tube. Surgeon and assistant stand on the right of the patient. A 10 mm camera port is placed 7th intercostals space in posterior axillary line, CO2 pneumothorax is created with pressure of 8mmHg. A 5 mm port is placed just posterior to the scapular tip. The last 10mm port is placed at 9th intercostals space in the scapular line for. The tumor and esophagus are dissected with cleaning of the lymph nodes along bilateral recurrent nerve.
  In controlling group, The four chest ports were similar to that described by the University of Pittsburgh group. The left two ports are used for surgical exposure, the right two ports is to divide and dissect the esophagus. The dissection is similar to that of the prone position.
  Other Names: MInimally invasive esophagectomy

SUMMARY:
The purpose of this prospective randomized study is to compare clinical outcomes from two different patient position(prone vs left decubitus)with thoracoscopic esophageal mobilization in the procedure of Minimally Invasive Esophagectomy (MIE).

* Comparing morbidities from the two groups
* Comparing short-term quality of life from the two groups
* Comparing oncological results (3,5 year survival) from the two groups

DETAILED DESCRIPTION:
Thoracoscopic esophagectomy is routinely performed in two positions. The left decubitus position is the most commonly used position at most centers. However prone position is another alternative.

The left decubitus position is advocated for its the same position as the open procedure and easy to learn, as well as easy to emergent conversion to open thoracotomy .However, the disadvantage of this position is the need of lung retraction for better exposure and definitely one lung ventilation. They are regarded as potential causes leading lung injury.

Prone thoracoscopic esophageal mobilization has been advocated for its potential benefits of increased operative exposure, no lung retraction, avoid one lung ventilation, improved surgeon ergonomics. But it is difficult to make emergent conversion under this positon and not familiar with most thoracic or digestive surgeons. A longer learning curve may be needed.

A few publications have compared the two position with thoracoscopic mobilization of the esophagus in retrospective study of a small cohort. Until now, no prospective randomized study has been carried out in this field.

ELIGIBILITY:
Inclusion Criteria:

* clinical stage I/II esophageal cancer
* normal blood test of basic metabolism panel
* pulmonary function: FEV1 > 1.2L, FEV1% > 50%, DLCO > 50%
* heart function: NY grade I and grade II
* sign informed consent

Exclusion Criteria:

* Patients who received neoadjuvant therapy
* Mental disorders

Ages: 35 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Estimated)
Dates: Start 2010-07; Primary Completion 2013-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Perioperative morbidity and mortality from the two groups | 1 -5 years after surgery

SECONDARY OUTCOMES:
short-term quality of life(postoperative 6 months and 1 year) between the two groups | 1 year
3-and 5-year survival rate between the two groups | 1 - 5 years after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Zhong Shan Hospital, Fu Dan University, Shanghai, China